CLINICAL TRIAL: NCT05751798
Title: A Multicenter, Phase 1/2, Dose-finding and Dose Expansion Study of OSE-279, a PD-1 Blocking Monoclonal Antibody, in Subjects With Advanced Solid Tumors or Lymphomas
Brief Title: Dose-finding and Dose Expansion Study of OSE-279 in Subjects With Advanced Solid Tumors or Lymphomas
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OSE Immunotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OSE-279-C101; 2022-001136-28 (EudraCT Number)
Record Dates: First submitted 2023-01-30; First posted 2023-03-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Solid Advanced Tumor; Lymphoma; NSCLC (Non-small Cell Lung Cancer)
Keywords: Solid advanced tumor; Lymphoma; Rare tumor; PD-L1 positive tumor; PD-1 blocking monoclonal antibody; NSCLC (non-small cell lung cancer); Cancer vaccine; Immune check point inhibitor
MeSH Terms: conditions — Lymphoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Part A: 3 dose levels: Dose selection (completed) Part B: 1 dose level: OSE-279 + OSE2101
  Note: Part C is conditional upon Part B. Part C: 2 dose levels s(HLA-A2 positive). 2:1 ratio: OSE-279 + OSE2101 or OSE-279.
  Part C: 1 dose level: OSE-279 (HLA-A2 negative)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A: OSE-279 100 mg (Experimental): Part A: Dose Level 1: OSE-279 100 mg
  Interventions: Drug: Part A: OSE-279 100mg
- Part A: OSE-279 300 mg (Experimental): Part A: Dose Level 2: OSE-279 300 mg
  Interventions: Drug: Part A: OSE-279 300mg
- Part A: OSE-279 600 mg (Experimental): Part A: Dose Level 3: OSE-279 600 mg
  Interventions: Drug: Part A: OSE-279 600mg
- Part B: OSE-279 600 mg and OSE2101 (Experimental): Part B: OSE-279 600 mg and OSE2101
  Interventions: Drug: Part B: OSE-279 600 mg and OSE2101
- Drug: Part C: OSE-279 600 mg and OSE2101 - HLA-A2 positif (Experimental): Part C: OSE-279 600 mg and OSE2101 - HLA-A2 positive
  Interventions: Drug: Part C: OSE-279 600 mg and OSE2101 - HLA-A2 positive
- Part C: OSE-279 600 mg - HLA-A2 positif (Experimental): Part C: OSE-279 600 mg - HLA-A2 positif
  Interventions: Drug: Part C: OSE-279 600 mg - HLA-A2 positif
- Part C: OSE-279 600 mg - HLA-A2 negative (Experimental): Part C: OSE-279 600 mg - HLA-A2 negative
  Interventions: Drug: Part C: OSE-279 600 mg - HLA-A2 negative

INTERVENTIONS:
Drug: Part A: OSE-279 100mg — Human IgG4 mAb against PD-1
  Arms: Part A: OSE-279 100 mg
Drug: Part A: OSE-279 300mg — Human IgG4 mAb against PD-1
  Arms: Part A: OSE-279 300 mg
Drug: Part A: OSE-279 600mg — Human IgG4 mAb against PD-1
  Arms: Part A: OSE-279 600 mg
Drug: Part B: OSE-279 600 mg and OSE2101 — OSE-279: OSE-279: Human IgG4 mAb against PD-1 OSE2101: Cancer vaccine
  Arms: Part B: OSE-279 600 mg and OSE2101
Drug: Part C: OSE-279 600 mg and OSE2101 - HLA-A2 positive — OSE-279: Human IgG4 mAb against PD-1 OSE2101: Cancer vaccine
  Arms: Drug: Part C: OSE-279 600 mg and OSE2101 - HLA-A2 positif
Drug: Part C: OSE-279 600 mg - HLA-A2 positif — OSE-279: Human IgG4 mAb against PD-1
  Arms: Part C: OSE-279 600 mg - HLA-A2 positif
Drug: Part C: OSE-279 600 mg - HLA-A2 negative — OSE-279: Human IgG4 mAb against PD-1
  Arms: Part C: OSE-279 600 mg - HLA-A2 negative

SUMMARY:
This is a phase 1/2, multicenter, dose-finding and dose expansion study of OSE-279, a PD-1 blocking monoclonal antibody, in subjects with advanced solid tumors or lymphomas.

DETAILED DESCRIPTION:
* The PART A objectives are to determine the Maximum Tolerated Dose (MTD) and/or the Recommended Phase 2 Doses (RP2D) when administered as single IV infusion on every 3 or 6 weeks.
* The PART B objective is to evaluate the safety of the combination of OSE-279 administered at the RP2D (600mg Q6W) and OSE2101 at the therapeutic dose as 1st line treatment of metastatic (stage IV) NSCLC.
* The PART C objective is to assess the antitumor activity of OSE-279 in combination with OSE2101 versus 0SE-279 in terms of overall response rate (ORR) as assessed locally, in patients with 1st line metastatic (stage IV) NSCLC.

ELIGIBILITY:
Parts B and C - INCLUSION CRITERIA

1. Male or female, aged ≥ 18 years
2. Signed and dated informed consent form (ICF) prior to any trialspecific procedures.
3. ECOG performance status 0-1
4. Patients must be affiliated to a social security system or an equivalent system, if applicable as per local regulations.
5. Patients expressing HLA-A2 phenotype on blood sample performed by an experienced laboratory using a validated test (PCR or NGS). Additional patients HLA-A2 negative will be included in PART C.
6. Tumor type: a) Histologically or cytologically documented Stage IV squamous or non-squamous NSCLC not eligible for definite surgery or radiation, without EGFR sensitizing mutation or ALK and ROS1 gene alterations eligible for targeted therapy or other mutations for which an approved therapy exists in 1st line metastatic (see protocol); b) PD-L1 expression by TPS ≥ 50% (local)
7. Patients with NO prior systemic therapy including immunotherapy in the first-line metastatic setting. In case of neoadjuvant/adjuvant therapy, therapy was completed at least 6 months prior to the diagnosis of metastatic disease.
8. Patients with at least one measurable lesion according to RECIST v1.1.
9. Adequate organ function:

   1. Bone marrow: neutrophils ≥ 1.5 x 109/L, hemoglobin ≥ 90 g/L, platelets ≥ 100 x 109/L
   2. Renal function: serum creatinine ≤ 1.5 ULN or CKDEPI creatinine clearance ≥ 30 mL/min
   3. Liver function: AST and ALT ≤ 3 ULN, bilirubin ≤ 1.5 ULN. In case of liver metastasis: AST and ALT ≤ 5 ULN. For patients with Gilbert's syndrome total bilirubin ≤ 3 ULN or direct bilirubin ≤ 1.5 ULN.

Parts B and C - NON-INCLUSION CRITERIA

1. Patient eligible to surgical resection or another approved therapeutic regimen known to provide clinical benefit; Known hypersensitivity to the active substances or to any of the excipients of OSE2101 or docetaxel.
2. Patient previously treated with approved/investigational anti-PD-1/PD-L1
3. Patient with active autoimmune disease or a documented history of autoimmune disease requiring systemic treatment (i.e., corticosteroids or immunosuppressive drugs); see exceptions in protocol
4. Patient participating in another clinical trial with a medicinal product
5. Patients who have not recovered from AEs (i.e. > G1 according to CTCAE v5.0) due to prior treatment with anti-cancer agents with exception of G2 neuropathy or any Grade alopecia. (see protocol)
6. Patients with known additional malignancy progressing or requiring active treatment. Basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer are not non-inclusion criteria
7. Patients with known active central nervous system metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to C1D1 and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids (at doses > 10 mg/day methylprednisolone or equivalent) for 4 weeks prior C1D1
8. Patients with active or history of non-infectious pneumonitis requiring steroids, or interstitial lung disease
9. Patients with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the duration of the study
10. Patients with a history of uncontrolled or symptomatic, clinically significant cardiovascular disease: stroke, myocardial infarction, angina pectoris, arrhythmias, congestive heart failure (NYHA Class >2), or myocarditis within 6 months prior to first study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Part A: Occurrence of dose limiting toxicity (DLT). Part B: Safety and tolerability of the combination OSE-279/OSE2101. Part C: Overall response rate (ORR) of the combination OSE-279/OSE2101 | Part A: DLT observation period is defined as the first 21 days after receiving the 1st injection of OSE-279 (Cycle 1) Part B: DLT observation period is defined as the first 6 weeks after receiving the combinaison Part C: Best response
  Part A: Occurrence of dose limiting toxicity (DLT) Part B: Occurrence of dose limiting toxicity (DLT) Part C: ORR: Complete Response (CR) and Partial Response (PR) rate

SECONDARY OUTCOMES:
Part A: Objective Response Rate (ORR). Part B: Complete Response (CR) and Partial Response (PR) rate. Part C: CR, PR and Stable Disease (SD) rate | Part A: Through study completion, an average of 1 year Part B: ORR, DCR, DOR, TTR, DCR at 12 weeks and 24 weeks, PFS, OS and OS at 12 months Part C: DCR,TTR, DOR, PFS at 12 weeks and 24 weeks, OS and OS rate at 12 months
  Part A: Objective Response Rate (ORR): complete response (CR) and partial response (PR), based on RECIST 1.1/RECIL and iRECIST Part B: Objective Response Rate (ORR): complete response (CR) and partial response (PR), based on RECIST 1.1/RECIL and iRECIST Part C: CR, PR and Stable Disease (SD) rate, based on RECIST 1.1/RECIL and iRECIST
Part A and Part B: Disease Control Rate (DCR: CR, PR and SD). Part C: Time to response | Part A: Through study completion, an average of 1 year
  Part A and Part B: Disease Control Rate (DCR): complete response (CR), partial response (PR) and stable disease (SD) based on RECIST 1.1/RECIL and iRECIST
Part A and Part B: Time to response. Part C: Duration of Objective Response (DOR) | Time
  Part A and Part B: Time to response
Part A and Part B: Duration of response (DR). Part C: Progression Free Survival (PFS) | Part A: From the first assessment of CR or PR until the date of the first occurrence of PD, or until the date of death (up to 1 year)
  Part A and Part B: Duration of response (DR). Part C: Progression Free Survival (PFS)
Part A and Part B: Progression Free Survival (PFS). Part C: DCR (CR+PR+SD) at 12 weeks and 24 weeks | Part A: From start of treatment until date of progression based on RECIST 1.1/RECIL and iRECIST or date of death (up to 1 year). Part C: DCR at 12 weeks and 24 weeks
  Part A and Part B: Progression Free Survival (PFS). Part C: DCR at 12 weeks and 24 weeks
Part A: DCR at 12 weeks (CR+PR+SD). Part B: DCR at 12 weeks and 24 weeks (CR+PR+SD). Part C: Overall Survival (OS) | Part A: Up to 12 weeks Part B: at 12 weeks and 24 weeks
  Part A: DCR at 12 weeks (CR+PR+SD). Part B: DCR at 12 weeks and 24 weeks (CR+PR+SD). Part C: Overall Survival.
Part A and Part B: Overall Survival (OS). Part C: Overall Survival (OS) rate. | Part A and Part C: From start of treatment to Death (up to 2 years). Part C: Overall Survival (OS) rate at 12 months.
  Part A and Part B: Overall Survival (OS). Part C: Overall Survival (OS) rate.
Part B: Overall Survival (OS) rate. | Part B: Overall Survival (OS) rate at 12months

CONTACTS AND LOCATIONS:
Locations (11):
- Belgium (2):
  - Institut Jules Bordet, Anderlecht
  - Antwerp University Hospital, Edegem
- France (6):
  - Centre Léon Bérard, Lyon
  - Hopital Saint Joseph, Paris
  - Centre Eugène Marquis, Rennes
  - Institut de Cancerologie de l'Ouest, Saint-Herblain
  - Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Spain (3):
  - University Hospital A Coruña Biomedical Research Institute (INIBIC), A Coruña
  - Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (IDIBGI), Girona
  - Hospital Regional Universitario de Málaga, Málaga

IPD SHARING:
Plan to Share IPD: Undecided